CLINICAL TRIAL: NCT01547650
Title: Evaluation of Plasma Volume Using Ultrasound in Disorders of Fluid With Sodium
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Nagaoka Red Cross Hospital (Other)
Responsible Party: Principal Investigator, Kyuzi Kamoi, Investigator, Nagaoka Red Cross Hospital
Other Study IDs: 3-Kamoi
Record Dates: First submitted 2012-02-23; First posted 2012-03-08 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2012-03

CONDITIONS: Other Diagnoses and Conditions

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — There is no biospeciment.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SIADH, CSWS, CDI, PP, DIH, HF: CSWS (cerebral salt wasting syndrome), SIADH (syndrome of inappropriate ADH) , CDI (central diabetes insipidus), PP (primary polydipsia), DIH (drug-induced hyponatremia), HF (heart failure with hyponatremia)
  Interventions: Other: Calculated CVP by using cardiac echogram

INTERVENTIONS:
Other: Calculated CVP by using cardiac echogram — Before and after the correction of plasma volume

SUMMARY:
Rossi NF & Schrier RW reported that for having differential diagnosis in hyponatremic state, it is important to have a grasp of extra cellular fluid (ECF) volume. However, recent works showed that it is not easy to estimate the ECF state using by physical findings and by usual laboratory methods.

Damaraju SC et al. first demonstrated that measuring central venous pressure (CVP) is significant to evaluate the ECF state in hyponatremic patients with intracranial diseases. Accordingly, it may be useful to measure the CVP in the hyponatremic patients. However, usually it is difficult to measure the CVP in all patients with hyponatremia because that the method is due to invasive procedure. With recently development, it is possible to estimate the CVP calculation using cardiac echogram without invasion. However, it is not clear that an evaluation by using such echogram estimates the state of ECF volume in hyponatremic patients.

Therefore, the investigators examine whether the CVP calculation by using cardiac echogram by Marcelino P et al. method without invasion is estimated such condition in hyponatremic patients before and after treatments.

As the primary endpoint, the VCI index values is investigated and compared with each group before and after correction of disorders of fluid with sodium. Furthermore, some variables including sodium, potassium, chloride, creatinine, BUN, uric acid, osmolality in blood and urine and plasma vasopressin are investigated and compared with each group before and after correction of disorders of fluid with sodium.

DETAILED DESCRIPTION:
Calculated CVP value as VCI (vena cava inferior) index by Marcelino P et al. method-they reported that VCI index using several echocardiographic parameters measured. A transthoracic echocardiographic study was performed using an Aloka SSD 2200 echocardiograph fitted with 2.5MHz probe with continuous-wave，pulsed and color Doppler (Japan). Using pulsed Doppler，each parameter is measured as following; the deceleration rime of E wave of tricuspid inflow，the gradient between right ventricle (RV) and right atrium (RA) by continuous Doppler，the VCI variation from the corresponding maximum expiratory diameter (measured at 2 cm from the RA and in dorsal decubitus) to its diameter during inspiration. All measurements were taken at the end-expiration in order to standardize the samples. VCI index = [tricuspid E deceleration (ms)] x 0.11 + [RV/RA gradient (mmHg)] x 0.16 - [VCI variation (mm)] (VCI, vena cava inferior; tricuspid E, tricuspid E wave; RV, right ventricle, RA, right atrium).

Na, Cl, K, creatinine, BUN and uric acid in serum and urine were measured by the usual methods before and after the correction of plasma volume. Further, osmolality and vasopressin in plasma and osmolality in urine were also measured by the usual methods.

ELIGIBILITY:
Inclusion Criteria:

Patients with disorders of fluid with sodium including cerebral salt wasting syndrome (CSWS), syndrome of inappropriate antidiuretic hormone secretion (SIADH), primary polydipsia (PP), central diabetes insipidus (CDI) and others

* Patients more than 18 years old (gender is disregarded)
* Healthy subjects more than 18 years old (gender is disregarded)

Exclusion Criteria:

Patients with a serious complication in the heart, liver or kidney

* Pregnant or possibly pregnant patients, or lactating patients
* Patients complicated with a malignant tumor at present.
* Patients participating in other clinical study.
* Other than the above, patients judged inappropriate as the subjects of this study by the investigator

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with disorders of fluid with sodium including cerebral salt wasting syndrome (CSWS), syndrome of inappropriate antidiuretic hormone secretion (SIADH), primary polydipsia (PP), central diabetes insipidus (CDI) and others
  * Patients more than 18 years old (gender is disregarded)
  * Healthy subjects more than 18 years old (gender is disregarded)
Sampling Method: Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2012-02; Primary Completion 2022-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Calculated CVP by using cardiac echogram | within the first 30 days (plus or minus 3 days) after correcting status of plasma volume

CONTACTS AND LOCATIONS:
Overall Officials: Kyuzi Kamoi, MD, Principal Investigator — Nagaoka Red Cross Hospital and University of Niigata Prefecture
Locations (1):
- Nagaoka Red Cross Hospital, Nagaoka, Niigata, Japan

REFERENCES:
- [Background] Damaraju SC, Rajshekhar V, Chandy MJ. Validation study of a central venous pressure-based protocol for the management of neurosurgical patients with hyponatremia and natriuresis. Neurosurgery. 1997 Feb;40(2):312-6; discussion 316-7. doi: 10.1097/00006123-199702000-00015. PMID 9007863